CLINICAL TRIAL: NCT05765331
Title: Evaluating the Effectiveness of Chatbot-Based Intervention on Enhancing Self-management and Decision Self-efficacy Among Men Having Lower Urinary Tract Symptoms With or Without Erectile Dysfunction in the Post COVID-19 Era
Brief Title: The Impact of Chatbot-aid on Promoting Self-management of Men's Health in the Post COVID-19 Era
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: (988)111A-66-2
Record Dates: First submitted 2023-03-05; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Benign Prostate Enlargement; Lower Urinary Tract Symptoms; Erectile Dysfunction
Keywords: Lower urinary tract symptoms; Erectile dysfunction; Men's Health; Chatbot; Chronic disease self-management; Decision self-efficacy
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot-aid intervention (Experimental): Chatbot-aid intervention group
  Interventions: Device: Chatbot
- Control group (No Intervention): Written routine nursing health education guidance intervention.

INTERVENTIONS:
Device: Chatbot — The AI chatbot is a kind of artificial intelligence technology that can help increase knowledge and understanding of men's health issues. That interacts with subjects through literal text and provides educational resources, advice, and assistance related to lifestyle changes. The chatbot is a valuable aid to increase men's health by providing information about enlarged prostate with urination problems and erectile dysfunction.
  Arms: Chatbot-aid intervention

SUMMARY:
The AI chatbot as an artificial intelligence technology provides disease information and health care through digital assistance. However, the effectiveness of chatbot in promoting men's health in the field of urology needs further research to evaluate its actual results. The purpose of this study is to explore the impact of AI chatbot-aid intervention on enhancing self-management, and decision self-efficacy among men with lower urinary tract symptoms (LUTS) due to an enlarged prostate, and with or without erectile dysfunction (ED) in the post COVID-19 era.

DETAILED DESCRIPTION:
1. Background and objectives :

   After the age of 50 years, men's health may be impacted by various disorders such as lower urinary tract symptoms (LUTS) and erectile dysfunction (ED). Due to a lack of understanding and awareness, patients often fail to recognize early signs and are not compliant with medical advice. As they are hesitant to discuss these issues related to urination and erectile functions, they avoid seeking medical help, especially due to the restrictions and concerns brought by the COVID-19 pandemic. Consequently, worsening symptoms can adversely affect their quality of life and dignity. Studies have found that providing men with self-management health programs results in better symptom management and medical decisions. Therefore, work is underway to develop artificial intelligence (AI) platforms to allow men to manage their health before consulting a doctor. Chatbots are used for various medical decisions and healthcare management, and can now provide men with various healthcare information to help improve the effectiveness of self-care and medical treatments in the post COVID-19 period.

   The purpose of this study is to explore the impact of AI chatbot aid intervention on enhancing self-management, and decision self-efficacy among men with lower urinary tract symptoms (LUTS) due to an enlarged prostate, with or without erectile dysfunction (ED) in the post COVID-19 era.
2. Materials and Methods:

2.1. Trial design and ethical approval

This was a 1:1 two groups randomized controlled trial (RCT) with pre- and post-test experimental design. This study was approved by the Institutional Review Board (IRB) of Cheng Hsin General Hospital in Taipei, Taiwan (approval number CHGH-IRB (988)111A-66-2) and participants were provided with informed consent. Both groups had similar demographics. One hundred male patients will be recruited from the Urology outpatient clinic, with 50 patients randomly assigned to the experimental group and 50 patients to the control group.

2.2 Participants

Patients diagnosed with health-related diseases by urologists were included in this study. The conditions were as follows:(1) male, (2) age between 45-80 years old, (3) prostate enlargement with lower urinary tract symptoms, (4) need a mobile phone and willing to download the line chatbot. The exclusion criterion was a history of psychosis.

2.3 Intervention

The study uses a chatbot in collaboration with the Taiwan Urological Association (TUA) and the Taiwan Continence Society (TCS), which is deployed on the line app for mobile devices. The chatbot uses an AI model integrated with the line developer platform to predict risks for men's health conditions such as urinary symptoms and erectile dysfunction. Patients can access the chatbot for free by scanning a QR code. It provides self-management advice on issues such as prostate enlargement, urinary symptoms, and erectile dysfunction. It also provides patient-centered decision-making aids that support and encourage patients, especially in improving urination and erectile dysfunction.

2.4 Research instruments

The patients in both groups were asked to complete a basic personal information form, as well as several questionnaires including the International Prostate Symptom Score (IPSS), International Index of Erectile Function-5 (IIEF-5), Men's Health knowledge score, Partners in Health (PIH), and Decision Self-Efficacy Scale (DSES) before and 2-4 weeks after receiving the intervention measures. Additional examination data, such as prostate-specific antigen (PSA), uroflowmetry, and prostate sonography, were collected from medical records. A satisfaction questionnaire was also administered to the patients.

2.5 Statistical methods

SPSS was used for statistical analysis, including McNemar's test and independent sample t-test were used to compare and analyze the difference in the knowledge score, self-management, and decision-making self-efficacy between the experimental group and control group before and after the intervention; paired t-test was used to compare individuals before and after receiving intervention measures; Pearson's correlation was used to analyze the relationship among LUTS, knowledge score, self-management, and decision self-efficacy; Finally, multiple regression analysis to analyze the impact of using the chatbot on satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 years to 80 years old
* Prostate enlargement with lower urinary tract symptoms
* Need a mobile phone and willing to download the line chatbot

Exclusion Criteria:

* Psychosis

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Men's Health Knowledge Score | Baseline and 2-4 weeks after intervention.
  The 15 items of the Men's Health knowledge score are based on urination, prostate, and erectile dysfunction disorders. A total of 6 domains are to create men's health knowledge, which is used to evaluate the effectiveness of chatbot in promoting men's health knowledge.
Partners in Health Scale | Baseline and 2-4 weeks after intervention.
  The Partners in Health (PIH) is a validated,12 items questionnaire scored on a self-rated 9-point Likert scale (range: 0-8; higher scores indicate better self-management).
Decision Self-Efficacy Scale | Baseline and 2-4 weeks after intervention.
  The 11 items of the Decision Self-Efficacy Scale (DSES) used to assess the self-confidence of participants in their ability to make health decisions, ranged from 0 (not at all confident) to 4 (very confident).

SECONDARY OUTCOMES:
The evaluation of chatbot satisfaction. | 2-4 weeks after intervention.
  There are 9 questions about the satisfaction level of using the chatbot, with a Likert scale of 1-5, where 1 is "extremely dissatisfied" and 5 is "extremely satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Kuo Chen, MD, PhD, Principal Investigator — Cheng-Hsin General Hospital
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Albarqouni L, Sanders S, Clark J, Tikkinen KAO, Glasziou P. Self-Management for Men With Lower Urinary Tract Symptoms: A Systematic Review and Meta-Analysis. Ann Fam Med. 2021 Mar-Apr;19(2):157-167. doi: 10.1370/afm.2609. PMID 33685877
- [Background] Barry MJ, Fowler FJ Jr, O'Leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT. The American Urological Association symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Association. J Urol. 1992 Nov;148(5):1549-57; discussion 1564. doi: 10.1016/s0022-5347(17)36966-5. PMID 1279218
- [Background] Blanker MH, Brandenbarg P, Slijkhuis BGC, Steffens MG, van Balken MR, Jellema P. Development of an online personalized self-management intervention for men with uncomplicated LUTS. Neurourol Urodyn. 2019 Aug;38(6):1685-1691. doi: 10.1002/nau.24040. Epub 2019 May 20. PMID 31107577
- [Background] Bortnick E, Brown C, Simma-Chiang V, Kaplan SA. Modern best practice in the management of benign prostatic hyperplasia in the elderly. Ther Adv Urol. 2020 May 27;12:1756287220929486. doi: 10.1177/1756287220929486. eCollection 2020 Jan-Dec. PMID 32547642
- [Background] Calogero AE, Burgio G, Condorelli RA, Cannarella R, La Vignera S. Epidemiology and risk factors of lower urinary tract symptoms/benign prostatic hyperplasia and erectile dysfunction. Aging Male. 2019 Mar;22(1):12-19. doi: 10.1080/13685538.2018.1434772. Epub 2018 Feb 2. PMID 29392976
- [Background] Capogrosso P, Boeri L, Pozzi E, Ventimiglia E, Schifano N, Abbate C, Matloob R, Deho F, Montorsi F, Salonia A. Is It Compulsory to Investigate for Erectile Dysfunction in Patients Presenting for Low Urinary Tract Symptoms? Eur Urol Focus. 2021 Jan;7(1):172-177. doi: 10.1016/j.euf.2019.08.007. Epub 2019 Aug 30. PMID 31474582
- [Background] Chapple C, Castro-Diaz D, Chuang YC, Lee KS, Liao L, Liu SP, Wang J, Yoo TK, Chu R, Sumarsono B. Prevalence of Lower Urinary Tract Symptoms in China, Taiwan, and South Korea: Results from a Cross-Sectional, Population-Based Study. Adv Ther. 2017 Aug;34(8):1953-1965. doi: 10.1007/s12325-017-0577-9. Epub 2017 Jul 7. PMID 28687936
- [Background] Dumbraveanu I, Ceban E, Banov P. Lower urinary tract symptoms and erectile dysfunction in men from the Republic of Moldova. J Med Life. 2018 Apr-Jun;11(2):153-159. PMID 30140322
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] Ghose A, Roy S, Vasdev N, Olsburgh J, Dasgupta P. The Emerging Role of Artificial Intelligence in the Fight Against COVID-19. Eur Urol. 2020 Dec;78(6):775-776. doi: 10.1016/j.eururo.2020.09.031. Epub 2020 Sep 17. PMID 32994064
- [Background] Goldenthal SB, Portney D, Steppe E, Ghani K, Ellimoottil C. Assessing the feasibility of a chatbot after ureteroscopy. Mhealth. 2019 Mar 15;5:8. doi: 10.21037/mhealth.2019.03.01. eCollection 2019. PMID 31019961
- [Background] Griffith JW, Messersmith EE, Gillespie BW, Wiseman JB, Flynn KE, Kirkali Z, Kusek JW, Bavendam T, Cella D, Kreder KJ, Nero JJ, Corona ME, Bradley CS, Kenton KS, Helfand BT, Merion RM, Weinfurt KP; LURN Study Group. Reasons for Seeking Clinical Care for Lower Urinary Tract Symptoms: A Mixed Methods Study. J Urol. 2018 Feb;199(2):528-535. doi: 10.1016/j.juro.2017.07.067. Epub 2017 Jul 20. PMID 28734864
- [Background] Li JO, Liu H, Ting DSJ, Jeon S, Chan RVP, Kim JE, Sim DA, Thomas PBM, Lin H, Chen Y, Sakomoto T, Loewenstein A, Lam DSC, Pasquale LR, Wong TY, Lam LA, Ting DSW. Digital technology, tele-medicine and artificial intelligence in ophthalmology: A global perspective. Prog Retin Eye Res. 2021 May;82:100900. doi: 10.1016/j.preteyeres.2020.100900. Epub 2020 Sep 6. PMID 32898686
- [Background] Nadarzynski T, Miles O, Cowie A, Ridge D. Acceptability of artificial intelligence (AI)-led chatbot services in healthcare: A mixed-methods study. Digit Health. 2019 Aug 21;5:2055207619871808. doi: 10.1177/2055207619871808. eCollection 2019 Jan-Dec. PMID 31467682
- [Background] Nadarzynski T, Puentes V, Pawlak I, Mendes T, Montgomery I, Bayley J, Ridge D. Barriers and facilitators to engagement with artificial intelligence (AI)-based chatbots for sexual and reproductive health advice: a qualitative analysis. Sex Health. 2021 Nov;18(5):385-393. doi: 10.1071/SH21123. PMID 34782055
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Wang TJ, Chiu PP, Chen KK, Hung LP. Efficacy of a decision support intervention for reducing decisional conflict in patients with elevated serum prostate-specific antigen: A randomized controlled trial. Eur J Oncol Nurs. 2021 Feb;50:101865. doi: 10.1016/j.ejon.2020.101865. Epub 2020 Nov 4. PMID 33212360
- See also: O'Connor, A. M. (2002). User manual-decisional self-efficacy scale. Ottawa: Ottawa Hospital Research Institute;1995 [modified 2002] — http://decisionaid.ohri.ca/docs/develop/user_manuals/UM_decision_selfefficacy.pdf